CLINICAL TRIAL: NCT05253898
Title: Comparison of Group-based Pelvic Floor Physical Therapy and Therapeutic Yoga for Postnatal Stress Urinary Incontinence
Brief Title: Comparison of Pelvic Floor Therapy and Yoga on Stres Urinary Incontinence Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Nergiz Sayın, Principal Investigator, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/005
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-01

CONDITIONS: Urinary Incontinence; Urinary Tract Disorders
Keywords: Urinary incontinence; Postnatal; Yoga; Pelvic floor muscle; Rehabilitation; Quality of life
MeSH Terms: conditions — Urinary Incontinence; Urologic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Floor Physical Therapy (Active Comparator): Group 1 includes a training program about correctly using pelvic floor muscles. At the first session, an educational program will be given to all women about the anatomy and function of the pelvic floor muscles. Then, the pelvic floor muscles contractions will be controlled by vaginal palpation for approximately 10 minutes.
  Then it will follow with 5 minutes of warm-up exercises, 30 minutes of fast and slow pelvic floor muscles contractions in different positions, and 10 minutes of abdominal breathing, general relaxation, stretching, and cool-down exercises.
  It is planned to teach contractions with internal palpation for 10 minutes before the first session to ensure that the patients' pelvic floor contractions are performed correctly. PFT treatment will be given as two sessions per week, 45 minutes, and 8 weeks as group sessions.
  Interventions: Procedure: Pelvic floor Physical Therapy
- Therapeutic Yoga Training (Active Comparator): Group 2 program includes therapeutic yoga training. It will begin with education about the positive effects of yoga on the body and pelvic floor.
  Then it will follow with 5 minutes of warm-up exercises, 30 minutes of different asanas coordinated with breathing, and 10 minutes of yogi breathing and cool-down exercises.
  Also, a home exercise program will be given based on yoga sessions. Participants will receive a detailed description of the home program.
  Interventions: Procedure: Therapeutic Yoga Training

INTERVENTIONS:
Procedure: Pelvic floor Physical Therapy — Purpose of pelvic floor muscle education program is reduce the symptoms of stress urinary incontinence and improving quality of life.
  Arms: Pelvic Floor Physical Therapy
Procedure: Therapeutic Yoga Training — Purpose of this group show the effectiveness of yoga therapy on stress urinary incontinence and quality of life.
  Arms: Therapeutic Yoga Training

SUMMARY:
The aim of this study is to compare the effectiveness of pelvic floor physical therapy (PFT) and therapeutic yoga training (TYT) for women who have postnatal stress urinary incontinence (SUI).

DETAILED DESCRIPTION:
32 subjects with postnatal stress urinary incontinence will be included in the study after a voluntary consent form will be filled out. Subjects will randomly be divided into two groups according to the order.

Pelvic floor physical therapy (PFT) (n=16) will be Group 1, and therapeutic yoga training (TYT) (n=16) will be the Group 2.

PFT group will be received sessions twice a week and a special home exercise program once a week for 8 weeks. Each session will include warm-up exercises, pelvic floor muscle contractions in different positions, and abdominal breathing techniques. Each session is planned for 45 minutes.

TYT group will be received sessions twice a week and a special home exercise program once a week for 8 weeks. Each session will include warm-up exercises, different asanas, and yogi breathing exercises. each session is planned for 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Women ages between 18 and 50 years old,
* Women who have SUI 45 days and above after giving birth
* Patients who accept to join the group sessions and will participate regularly in the treatment program

Exclusion Criteria:

* Women who have pelvic organ prolapsus and fecal incontinence
* Women who have undergone surgery for the lower urinary system
* Those who receive medication treatment for incontinence in the last 3 months
* Those with acute infection and bladder stones or tumors will not be included in the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 32 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-06-13 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
İncontinence Questionary at 8 weeks | Change from Baseline in incontinence questionary at 8 weeks
  İncontinence Questionary-3 (3IQ) is a simple questionnaire to categorize the type of urinary incontinence.
  First question evaluates the existence of incontinence in the past 3 months. Second and third questions are directed to familiarity and the existence of the types of incontinence.
  The 3IQ is a quick test to evaluate the types of urinary incontinence with high sensitivity especially for stress urinary incontinence.
Incontinence Severity Index | Change from Baseline in Incontinence Severity Index at 8 weeks
  Incontinence Severity Index (ISI) is a tool for assessing the severity of female urinary incontinence. ISI is consists of 2 questions to establish frequency and amount of leakage. The results categorize the severity into 4 as; slight, moderate, severe, and very severe.
Incontinence Quality of Life | Change from Baseline in Incontinence Quality of Life at 8 weeks
  Incontinence Quality of Life (I-QoL) is used for assessing the decrease of quality of life depending on urinary incontinence symptoms. I-QoL consists of 22 questions and results with 4 domains. I-QoL has identified the 3 factors; avoidance and limiting behavior (8 items), psychosocial impacts (9 items), and social embarrassment (5 items).
Global Perception of Improvement | Change from Baseline in Global Perception of Improvement at 8 weeks
  Global Perception of Improvement (GPI) is used for showing the individual improvement of healing depending patient's perspective. GPI is rated to the satisfaction of advancement depending on the treatment for patients. Patients rated themselves as much better, better, about the same, worse, and much worse.
Pelvic Floor Muscle Strength assessing with PERFECT | Change from Baseline in PERFECT degrees at 8 weeks
  PERFECT is used to assess pelvic floor muscle power, endurance, maximal repetitions, and the number of fast contractions by using internal digital palpation.
  (P) symbolizes the power and this value is identified with modified oxford Scale during max. volunteer contraction.
  (E) symbolizes the endurance and it's identified by how much time will continue the max. volunteer contraction.
  (R) symbolizes the repetitions and it's identified with the number of maximum volunteer contractions, between each contraction, must be 4 s resting time.
  (F) symbolizes the fast and it's identified the number of fast contractions.
  (ECT) symbolizes every contraction time which means recording all numbers and times during evaluation.
1 hour Pad Test | Change from Baseline in Pad Test at 8 weeks
  Pad test is an objective way to scale the amount of incontinence in a specific time and the same conditions. The test begins with drinking 500ml water and 30 minutes sitting, then equal repetitions of jumping, walking, coughing, bending down, and washing hands-on running water for each patient.
State-Trait Anxiety Inventory | Change from Baseline in State-Trait Anxiety Inventory at 8 weeks
  State-Trait Anxiety Inventory (STAI) form consist of 2 different tool. STAI-I examines the current anxiety level, and STAI-II examines the aspects of anxiety proneness general states of calmness and confidence. STAI-I consist of 20 questions about how person feel during the test. STAI-II consist of 20 questions about continues anxiety level.
Bladder Diary | Change from Baseline in Bladder Diary at 8 weeks
  Bladder diary is used to asses lower urinary tract symptoms (LUTS).

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur Tuncer, PT, PhD, Study Director — Hasan Kalyoncu University
Locations (1):
- Special Nova Therapy and Rehabilitation Center, Diyarbakır, Turkey (Türkiye)

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322